CLINICAL TRIAL: NCT00527150
Title: A Phase 1, Investigator And Subject Blind (Sponsor Open), Randomized, Placebo Controlled, Parallel Group, Multiple Dose Escalation Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Varenicline Amt-8 Controlled Release Formulation In Adult Smokers
Brief Title: Multiple Dose, Dose Escalation Study of Varenicline Controlled Release Formulation in Adult Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051069
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Other): Subjects will be randomized to receive either experimental drug (N=9) or matching placebo (N=3).
  Interventions: Drug: Varenicline Tartrate
- Cohort 2 (Other): Subjects will be randomized to receive either experimental drug (N=9) or matching placebo (N=3).
  Interventions: Drug: Varenicline Tartrate
- Cohort 3 (Other): Subjects will be randomized to receive either experimental drug (N=9) or matching placebo (N=3).
  Interventions: Drug: Varenicline Tartrate
- Optional Cohort 4 (Other): Subjects will be randomized to receive either experimental drug (N=9) or matching placebo (N=3).
  Interventions: Drug: Varenicline Tartrate
- Optional Cohort 5 (Other): Subjects will be randomized to receive either experimental drug (N=9) or matching placebo (N=3).
  Interventions: Drug: Varenicline Tartrate

INTERVENTIONS:
Drug: Varenicline Tartrate — Varenicline 1.8 mg AMT-8 controlled release tablets administered twice a day for 14 days.
  Arms: Cohort 1
Drug: Varenicline Tartrate — Planned dose is Varenicline 2.4 mg AMT-8 controlled release tablets administered twice a day for 14 days. Actual dose may be adjusted based on emerging data from prior dose cohorts.
  Arms: Cohort 2
Drug: Varenicline Tartrate — Planned dose is Varenicline 3 mg AMT-8 controlled release tablets administered twice a day for 14 days. Actual dose may be adjusted based on emerging data from prior dose cohorts.
  Arms: Cohort 3
Drug: Varenicline Tartrate — The dose to be administered is not yet determined and will be based on emerging data from prior dose cohorts. The dose will be administered as Varenicline AMT-8 controlled release tablets twice a day for 14 days. The doses to be tested may be lower, higher or repeat a previously tested dose and may include a titration.
  Arms: Optional Cohort 4
Drug: Varenicline Tartrate — The dose to be administered is not yet determined and will be based on emerging data from prior dose cohorts. The dose will be administered as Varenicline AMT-8 controlled release tablets twice a day for 14 days. The doses to be tested may be lower, higher or repeat a previously tested dose and may include a titration.
  Arms: Optional Cohort 5

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of escalating multiple oral doses of varenicline AMT 8 controlled release formulation for 14 days in adult smokers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.
* Currently smoking and have smoked an average of at least 10 cigarettes per day during the past year, with no period of abstinence greater than 3 continuous months in the past year.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Pregnant or nursing women are excluded; women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception as outlined in the protocol from at least 14 days prior to study medication administration until completion of protocol-required procedures are excluded.
* Subjects with an estimated creatinine clearance (CLcr) <80 mL/min derived using the method of Cockcroft and Gault.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic endpoints include varenicline area under the curve from 0-24 hours (AUC24), maximum plasma concentration (Cmax), | Day 1 and Day 14
Safety endpoints include evaluation of clinical safety laboratory tests, supine vital signs, triplicate 12-lead ECGs and adverse events. | up to 14 days
Time of maximum plasma concentration (Tmax) on Day 1 and Day 14 | Day 1 and Day 14
Minimum plasma concentration (Cmin), terminal half life (t1/2), observed accumulation ratio (Rac), peak:trough fluctuation (%PTF) on Day 14 only. | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, East Grand Forks, Minnesota
  - Pfizer Investigational Site, Fargo, North Dakota

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051069&StudyName=Multiple%20Dose%2C%20Dose%20Escalation%20Study%20of%20Varenicline%20Controlled%20Release%20Formulation%20in%20Adult%20Smokers